CLINICAL TRIAL: NCT03554486
Title: Evaluation of Fiasp® (Fast Acting Insulin Aspart) in 670G Hybrid Closed-Loop Therapy: To Assess How the 670G System Adapts to the Introduction of Fiasp® Insulin
Brief Title: Evaluation of Fiasp® (Fast Acting Insulin Aspart) in 670G Hybrid Closed-Loop Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Bruce Buckingham, Professor of Pediatric Endocrinology, Stanford University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 46202
Record Dates: First submitted 2018-05-31; First posted 2018-06-13 (Actual); Results first posted 2021-08-18 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Aspart

STUDY DESIGN:
Intervention Model Description: Subjects will be randomly assigned to start with either Fiasp insulin or Novolog insulin. After 2 weeks, they will start the previously unassigned insulin and continue using it for another 2 weeks.
Who Masked: Participant, Investigator
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fiasp then Novolog (Experimental): Following a 2-week run-in period for pump-setting adjustments and monitoring, participants 1 will use Fiasp insulin for 2 weeks, followed by Novolog insulin for 2 weeks. Both the subject and the investigator will be blinded to which group the subject is assigned.
  Interventions: Drug: Fiasp; Drug: Novolog
- Novolog then Fiasp (Experimental): Following a 2-week run-in period for pump-setting adjustments and monitoring, participants 1 will use Novolog insulin for 2 weeks, followed by Fiasp insulin for 2 weeks. Both the subject and the investigator will be blinded to which group the subject is assigned.
  Interventions: Drug: Fiasp; Drug: Novolog

INTERVENTIONS:
Drug: Fiasp — Fiasp insulin will be used for 2 weeks with the 670G hybrid closed-loop system
  Other Names: Fast Acting Insulin Aspart
Drug: Novolog — Novolog insulin will be used for 2 weeks with the 670G hybrid closed-loop system
  Other Names: Insulin Aspart

SUMMARY:
This is a pilot outpatient study conducted at Stanford to obtain preliminary data on how Fiasp® works in a closed-loop system and to determine if any changes need to be made to the 670G pump to optimize the use of Fiasp®.

DETAILED DESCRIPTION:
This will be a randomized cross-over blinded study and to see how the 670G pump responds to the introduction of Fiasp® insulin. Subjects enrolled in the study will have a 2 week period of optimization with weekly assessments of their Carelink download before entering the blinded phase of the study. They will use their usual home insulin during the optimization phase. They will then be started on their first blinded insulin (aspart or Fiasp®) which they will use for 2 weeks, before they cross-over to the other insulin.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of type 1 diabetes and using 670G pump for at least 1 month, and willing to have the 670G pump downloaded into a Carelink Clinical research database.
2. The diagnosis of type 1 diabetes is based on the investigator's judgment; C-peptide level and antibody determinations are not needed.
3. Age ≥18 years
4. Using Novolog or Fiasp® insulin at time of enrollment
5. Willing to use Fiasp® insulin
6. Total daily insulin dose is at least 0.3 units/kg/day
7. Usual carbohydrate intake is at least 60 grams a day, and willing to have at least 25 grams of carbohydrates for breakfast
8. For females, not currently known to be pregnant
9. An understanding of and willingness to follow the protocol and sign the informed consent
10. Willing to have photographs taken of their infusion sites
11. Willing to download their 670G pump every 1-2 weeks to a research Carelink account
12. Willingness to answer a brief online questionnaire every 2 weeks
13. Must be able to understand spoken or written English
14. For subjects participating in Part 2 of this study they will need to be using Fiasp® as part of their usual care
15. Hemoglobin A1c between 6 and 10% at the time of enrollment

Exclusion Criteria:

1. Pregnant or lactating females
2. No hypoglycemic seizure or loss of consciousness in the past 6 months
3. Severe episode of DKA in the 6 months prior to study enrollment that was unrelated to an infusion set failure
4. No known cardiovascular events in the last 6 months
5. No active proliferative diabetic retinopathy
6. Known tape allergies
7. Current treatment for a seizure disorder
8. Cystic fibrosis
9. Active infection
10. A known medical condition that in the judgment of the investigator might interfere with the completion of the protocol
11. Inpatient psychiatric treatment in the past 6 months
12. Presence of a known adrenal disorder
13. If on antihypertensive, thyroid, anti-depressant or lipid lowering medication, with lack of stability on the medication for the past 2 months prior to enrollment in the study
14. Abuse of alcohol
15. Dialysis or renal failure
16. Known eGFR <60%

Note: Adequately treated thyroid disease and celiac disease do not exclude subjects from enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-07-23 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Buckingham, MD, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Stanford University, Palo Alto, California
  - Stanford, Palo Alto, California

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zijlstra E, Demissie M, Graungaard T, Heise T, Nosek L, Bode B. Investigation of Pump Compatibility of Fast-Acting Insulin Aspart in Subjects With Type 1 Diabetes. J Diabetes Sci Technol. 2018 Jan;12(1):145-151. doi: 10.1177/1932296817730375. Epub 2017 Sep 18. PMID 28918652
- [Background] Bode BW, Johnson JA, Hyveled L, Tamer SC, Demissie M. Improved Postprandial Glycemic Control with Faster-Acting Insulin Aspart in Patients with Type 1 Diabetes Using Continuous Subcutaneous Insulin Infusion. Diabetes Technol Ther. 2017 Jan;19(1):25-33. doi: 10.1089/dia.2016.0350. Epub 2017 Jan 5. PMID 28055230
- [Background] Hsu L, Buckingham B, Basina M, Ekhlaspour L, von Eyben R, Wang J, Lal RA. Fast-Acting Insulin Aspart Use with the MiniMedTM 670G System. Diabetes Technol Ther. 2021 Jan;23(1):1-7. doi: 10.1089/dia.2020.0083. PMID 32520594

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 27 participants signed informed consent. 3 participants failed screening and did not enter the run-in period (a 2-week period for pump-setting adjustments and monitoring).
Groups:
- All Participants (run-in Period): Participants entered a 2-week run-in period prior to randomization.
- Fiasp Then Novolog: Following randomization after a 2-week run-in period, participants use Fiasp insulin for 2 weeks, followed by Novolog insulin for 2 weeks.
- Novolog Then Fiasp: Following randomization after a 2-week run-in period, participants use Novolog insulin for 2 weeks, followed by Fiasp insulin for 2 weeks.
Period: Run-in Period (2 Weeks)
Arm/Group | All Participants (run-in Period) | Fiasp Then Novolog | Novolog Then Fiasp
Started | 24 | 0 | 0
Completed | 21 | 0 | 0
Not Completed | 3 | 0 | 0
Not completed — Need for steroid injection | 1 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0
Period: Treatment Period 1 (2 Weeks)
Arm/Group | All Participants (run-in Period) | Fiasp Then Novolog | Novolog Then Fiasp
Started | 0 | 11 | 10
Completed | 0 | 10 | 9
Not Completed | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 1
Period: Treatment Period 2 (2 Weeks)
Arm/Group | All Participants (run-in Period) | Fiasp Then Novolog | Novolog Then Fiasp
Started | 0 | 10 | 9
Completed | 0 | 10 | 9
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants who completed the protocol are included in the analysis.
Groups:
- Fiasp Then Novolog: Following a 2-week run-in period, participants use Fiasp insulin for 2 weeks, followed by Novolog insulin for 2 weeks.
- Novolog Then Fiasp: Following a 2-week run-in period, participants use Novolog insulin for 2 weeks, followed by Fiasp insulin for 2 weeks.
- Total: Total of all reporting groups
Arm/Group | Fiasp Then Novolog | Novolog Then Fiasp | Total
Number analyzed (Participants) | 10 | 9 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.0 (15.2) | 44.1 (20.4) | 40.4 (17.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 9
  Male | 4 | 6 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 9 | 9 | 18
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 9 | 9 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 9 | 19
Hemoglobin A1C [Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin] | 7.1 (0.9) | 7.1 (0.5) | 7.1 (0.7)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Time in Range: Sensor Glucose Values Between 70-180 mg/dl
Description: Measured as percentage of time in range (days).
Time Frame: 7 days (during 2nd half of 2-week intervention period)
Population: Participants who completed the protocol are included in the analysis.
Measure: Mean (Standard Deviation); unit: percentage of time
Groups:
- Fiasp Insulin: Participants use Fiasp insulin for 2 weeks.
- Novolog Insulin: Participants use Novolog insulin for 2 weeks.
Arm/Group | Fiasp Insulin | Novolog Insulin
Number analyzed (Participants) | 19 | 19
percentage of time | 78.4 (9.3) | 75.3 (9.5)
Statistical Analysis 1: Comparison: Fiasp Insulin vs Novolog Insulin; Test type: Other; p = 0.051, t-test, 2 sided

2. Primary Outcome: Percentage of Time in Range: Sensor Glucose Readings <70 mg/dl
Description: Percentage of time in range (days) as a measure of hypoglycemia.
Time Frame: 7 days (during 2nd half of 2-week intervention period)
Population: Participants who completed the protocol are included in the analysis.
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Fiasp Insulin | Novolog Insulin
Number analyzed (Participants) | 19 | 19
percentage of time | 2.3 (2.0) | 3.1 (2.1)
Statistical Analysis 1: Comparison: Fiasp Insulin vs Novolog Insulin; Test type: Other; p = 0.17, t-test, 2 sided

3. Secondary Outcome: Mean Sensor Glucose in mg/dl
Description: Mean sensor data over the second week of using a randomized, blinded insulin.
Time Frame: 7 days (during 2nd half of 2-week intervention period)
Population: Participants who completed the protocol are included in the analysis.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Fiasp Insulin | Novolog Insulin
Number analyzed (Participants) | 19 | 19
mg/dL | 146 (12) | 147 (12)
Statistical Analysis 1: Comparison: Fiasp Insulin vs Novolog Insulin; Test type: Other; p = 0.74, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 6 weeks
Groups:
- Run-in Period: Participants with events occurring prior to randomization.
- Fiasp Insulin: Participants with events occurring during Fiasp insulin treatment.
- Novolog Insulin: Participants with events occurring during Novolog insulin treatment.
Arm/Group | Run-in Period | Fiasp Insulin | Novolog Insulin
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/19 | 1/19
Other Adverse Events (participants affected / at risk) | 0/28 | 0/19 | 1/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Run-in Period (N=28) | Fiasp Insulin (N=19) | Novolog Insulin (N=19)
Infusion set failure (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Run-in Period (N=28) | Fiasp Insulin (N=19) | Novolog Insulin (N=19)
Irritation/Inflammation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-30): https://cdn.clinicaltrials.gov/large-docs/86/NCT03554486/Prot_SAP_000.pdf